CLINICAL TRIAL: NCT00377910
Title: Placebo Controlled Trial, Testing the Efficacy of Polidocanol Injections as a Treatment of Chronic Achilles Tendinopathy.
Brief Title: The Efficacy of Polidocanol Injections as a Treatment of Chronic Achilles. Tendinopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: ON-02-012-OSi
Record Dates: First submitted 2006-09-18; First posted 2006-09-19 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Achilles Tendinopathy
Keywords: Chronic Achilles tendinopathy; Polidocanol; Ultrasound; Efficacy; RCT
MeSH Terms: interventions — Polidocanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1, drug (Active Comparator): Injections of polidocanol
  Interventions: Drug: Aethoxysclerol
- 2 drug (Placebo Comparator): injections of lidocaine
  Interventions: Drug: Aethoxysclerol

INTERVENTIONS:
Drug: Aethoxysclerol — 2 ml Aethoxysclerol 10 mg/ml 2 ml. lidocaine 10mg/ml
  Other Names: 1. drug: Polidocanol; 2. drug: Lidocaine

SUMMARY:
Chronic achilles tendinopathy is a common disease especially in adults. The golden standard in treatment has up to now been excentric exercises but with varying success. A new hypothesis is that this chronic pain is due to neo vascularisation. In a pilot study sclerosing injections with polidocanol have had a successful efficacy. Our aim is to study the efficacy of polidocanol as a treatment in a randomised controlled setting on a larger scale.

DETAILED DESCRIPTION:
48 patients with chronic achilles tendinopathy for more than 3 months who have tried excentric exercises without success will be randomised to either polidocanol or lidocaine injections if having ultrasound verified neo-vascularisation.

ELIGIBILITY:
Inclusion Criteria:

* 18 year old, Ultrasound verified Achilles tendinopathy with neo-vascularisation, pain duration more than three months, excentric exercises for at least three months, women: negative pregnancy test, safe anticonceptive

Exclusion Criteria:

* Dementia, mental disease or other illness incompatible with participation, no ultrasound verified neo-vascularisation, any illness which contraindicate the use of Polidocanol or Lidocaine, granulation tissue of more than 50 % of the Achilles tendon, ability of lying in prone position, women: pregnancy or breastfeeding,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Pain during physical activity which usually causes pain | 3 and 6 months

SECONDARY OUTCOMES:
Achilles tendon pressure measuring until pain release. | 3 and 6 months
Pain while resting. | 3 and 6 months
Patient evaluation of treatment efficacy | 3 and 6 months
FAOS | 3 and 6 months
AOFAS | 3 and 6 months
Number of neo-vascularisation. | day 0, 1 and 3 months
Localisation of the neo-vascularisation | day 0, 1 and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ole Simonsen, MD, DMSci, Principal Investigator — Northern Orthopaedic Division, Denmark
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

REFERENCES:
- [Background] Alfredson H, Ohberg L. Sclerosing injections to areas of neo-vascularisation reduce pain in chronic Achilles tendinopathy: a double-blind randomised controlled trial. Knee Surg Sports Traumatol Arthrosc. 2005 May;13(4):338-44. doi: 10.1007/s00167-004-0585-6. Epub 2005 Feb 2. PMID 15688235